CLINICAL TRIAL: NCT02121652
Title: Translating CBT-Insomnia for Lung Cancer Into Practice: A RCT
Brief Title: Cognitive Behavioral Therapy (CBT)-Insomnia for Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Suzanne Dickerson, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 517176-3; 517176-1 (Registry Identifier: SUNY UB IRB); 1R15NR013779-01A1 (NIH)
Record Dates: First submitted 2013-10-25; First posted 2014-04-23 (Estimated); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Chronic Insomnia
Keywords: lung cancer survivors; insomnia treatment; cognitive behavioral therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy eating control (Active Comparator): Healthy eating control involves healthy eating content delivered in a 90 minute group session with two follow up phone calls.
  Interventions: Behavioral: Healthy eating control
- Cognitive behavioral therapy (Experimental): Cognitive behavioral therapy for insomnia includes content on sleep restriction, stimulus control, relaxation, cognitive restructuring and sleep hygiene content delivered in a 90 minute group intervention with two follow up phone calls.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia — Cognitive behavioral therapy for insomnia includes content on sleep restriction, stimulus control, relaxation, cognitive restructuring and sleep hygiene content delivered in a 90 minute group intervention with two follow up phone calls.
  Arms: Cognitive behavioral therapy
Behavioral: Healthy eating control — Healthy eating control involves healthy eating content delivered in a 90 minute group session with two follow up phone calls.
  Arms: Healthy eating control

SUMMARY:
The purpose of this study is to determine whether cognitive behavioral therapy (CBT) is effective for insomnia in lung cancer survivors.

DETAILED DESCRIPTION:
A randomized controlled clinical trial will be used to test the efficacy of this brief CBT-I compared to attention control on sleep, mood, functional status and quality of life in lung cancer survivors and evaluate the feasibility of translating an evidence-based CBT-I into the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* 6 weeks from surgery for stage 1 or 2 Non Small Cell Lung Cancer
* chronic insomnia

Exclusion Criteria:

* Other preexisting sleep disorders
* Unstable medical illnesses

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Dickerson, RN, PhD, Principal Investigator — SUNY University at Buffalo School of Nursing
Locations (2):
- United States (2):
  - SUNY University at Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute Thoracic Clinic, Buffalo, New York

IPD SHARING:
Plan to Share IPD: Yes
Data have been prepared for sharing with other investigators. All collected individual participant data (IPD) can be accessed at our data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available one year after publication of the study findings manuscript.
Access Criteria: IPD will be publicly available to the public via a data repository.

REFERENCES:
- [Background] Edinger JD, Wohlgemuth WK, Radtke RA, Coffman CJ, Carney CE. Dose-response effects of cognitive-behavioral insomnia therapy: a randomized clinical trial. Sleep. 2007 Feb;30(2):203-12. doi: 10.1093/sleep/30.2.203. PMID 17326546
- [Background] Edinger JD, Sampson WS. A primary care "friendly" cognitive behavioral insomnia therapy. Sleep. 2003 Mar 15;26(2):177-82. doi: 10.1093/sleep/26.2.177. PMID 12683477
- [Background] Germain A, Shear MK, Hall M, Buysse DJ. Effects of a brief behavioral treatment for PTSD-related sleep disturbances: a pilot study. Behav Res Ther. 2007 Mar;45(3):627-32. doi: 10.1016/j.brat.2006.04.009. Epub 2006 Jun 14. PMID 16777060
- [Background] Espie CA, Fleming L, Cassidy J, Samuel L, Taylor LM, White CA, Douglas NJ, Engleman HM, Kelly HL, Paul J. Randomized controlled clinical effectiveness trial of cognitive behavior therapy compared with treatment as usual for persistent insomnia in patients with cancer. J Clin Oncol. 2008 Oct 1;26(28):4651-8. doi: 10.1200/JCO.2007.13.9006. Epub 2008 Jun 30. PMID 18591549
- [Background] Vena C, Parker K, Allen R, Bliwise D, Jain S, Kimble L. Sleep-wake disturbances and quality of life in patients with advanced lung cancer. Oncol Nurs Forum. 2006 Jul 1;33(4):761-9. doi: 10.1188/06.ONF.761-769. PMID 16858458
- [Background] Davidson JR, Feldman-Stewart D, Brennenstuhl S, Ram S. How to provide insomnia interventions to people with cancer: insights from patients. Psychooncology. 2007 Nov;16(11):1028-38. doi: 10.1002/pon.1183. PMID 17352006
- [Background] Dean GE, Redeker NS, Wang YJ, Rogers AE, Dickerson SS, Steinbrenner LM, Gooneratne NS. Sleep, mood, and quality of life in patients receiving treatment for lung cancer. Oncol Nurs Forum. 2013 Sep;40(5):441-51. doi: 10.1188/13.ONF.441-451. PMID 23989018
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Dean GE, Weiss C, Jungquist CR, Klimpt ML, Alameri R, Ziegler PA, Steinbrenner LM, Dexter EU, Dhillon SS, Lucke JF, Dickerson SS. Nurse-Delivered Brief Behavioral Treatment for Insomnia in Lung Cancer Survivors: A Pilot RCT. Behav Sleep Med. 2020 Nov-Dec;18(6):774-786. doi: 10.1080/15402002.2019.1685523. Epub 2019 Oct 31. PMID 31672070

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four participants were excluded from the study after screening positive (e.g. > or = to 15) on the overnight ApneaLink test and referred to sleep medicine for further assessment.
Period: Overall Study
Arm/Group | Healthy Eating Control | Cognitive Behavioral Therapy
Started | 20 | 20
Completed | 14 | 16
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Cognitve Behaviroal Therapy: Cognitive behavioral therapy for insomnia includes content on sleep restriction, stimulus control, relaxation, cognitive restructuring and sleep hygiene content delivered in a 90 minute group intervention with two follow up phone calls.
  Cognitive behavioral therapy for insomnia: Cognitive behavioral therapy for insomnia includes content on sleep restriction, stimulus control, relaxation, cognitive restructuring and sleep hygiene content delivered in a 90 minute group intervention with two follow up phone calls.
- Total: Total of all reporting groups
Arm/Group | Healthy Eating Control | Cognitve Behaviroal Therapy | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Mean (Standard Deviation); unit: years] | 64.45 (8.00) | 66.45 (7.51) | 65.45 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency
Description: Sleep Efficiency > 85% measured with a seven-day sleep diary. The score is calculated based on participants' recording of time asleep (minutes) divided by time in bed (minutes).
  Sleep Efficiency greater than or equal to 85% indicates good sleep quality, and values less than 85% indicate poor sleep quality.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: percentage of sleep efficiency
Groups:
- Healthy Eating Control: Healthy Eating Control
- Cognitive Behavioral Therapy: Cognitive Behavioral Therapy
Arm/Group | Healthy Eating Control | Cognitive Behavioral Therapy
Number analyzed (Participants) | 11 | 14
percentage of sleep efficiency | 79.70 (10.21) | 85.21 (20.54)

ADVERSE EVENTS:
Time Frame: one month
Description: Daytime Sleepiness
Arm/Group | Healthy Eating Control | Cognitve Behaviroal Therapy
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14
Other Adverse Events (participants affected / at risk) | 0/11 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes